CLINICAL TRIAL: NCT04959825
Title: Effect of Preoperative Melatonin in Inhaled Anesthetic Consumption
Brief Title: The Role of Preoperative Melatonin in Reducing the Inhaled Isoflurane Requirements in Open Nephrectomy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amany Hassan Saleh, Associate professor of anesthesia, surgical intensive care and pain management, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: MD-249-2020
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be allocated to the study groups using a computer-generated random list, and the group assignments will be sealed in sequentially numbered opaque envelopes that will be opened before induction of anesthesia. The data collector will be blinded to the group assignment and to the monitoring anesthetist, and the person who will give the drug will not bethe data collector.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- melatonin group (Active Comparator): Melatonin group (group M )will receive melatonin as a premedication 1 hour before surgery in a dose of 5 mg
  Interventions: Drug: Melatonin 5 mg
- control group (Placebo Comparator): 15 patients will be enrolled for open nephrectomy will receive sugar-coated tablets. Control group(group C)
  Interventions: Drug: Sugar Coated Tablets

INTERVENTIONS:
Drug: Melatonin 5 mg — study the effect of preoperative oral melatonin 5mg on isoflurane consumption and postoperative pain
  Arms: melatonin group
Drug: Sugar Coated Tablets — the control group patients will receive placebo tablets one hour before induction of anesthesia
  Arms: control group

SUMMARY:
Melatonin is a hormone that the pineal gland in the brain produces. Melatonin fulfills many functions in the body but it is mostly known for maintaining a circadian rhythm that is governed by the central circadian pacemaker (biological clock) in the suprachiasmatic nuclei in the hypothalamus. Melatonin works by attaching to receptors or nerve endings in the suprachiasmatic nucleus (SCN) in the hypothalamus. It binds to melatonin receptor 1 and melatonin receptor 2, commonly referred to as MT1 and MT2. People can take it as a natural or synthetic supplement to promote restful sleep. Melatonin showed promise for preventing shifts in sleep and wake times in people with jetlag and improving sleep in people with insomnia. It can also be used for headaches, cancer, and Alzheimer's disease.

Melatonin can be used as an analgesic, sedative, and hypnotic drug that can distinguish it as an attractive alternative premedicant

DETAILED DESCRIPTION:
A study that was done before in J Anaesth by Borazan H et al revealed that postoperative pain score in patients undergoing radical prostatectomy who received melatonin one hour before surgery as a premedication was significantly lower than the control group with a significant P-value( less than 0.05).

The entropy is indicated for adult and pediatric patients older than 2 years intraoperatively for monitoring the electric state of the brain. In adult patients, state entropy and response entropy can be used as an aid in monitoring the effects of certain anaesthetic agents which will help the user to titrate the anaesthetic agent according to the individual needs of each patient.

Furthermore, the use of entropy parameters may be associated with a reduction of anaesthetic use and faster emergence of anaesthesia. The entropy measurement is to be used as an adjunct to other physiological parameters.

To the best of investigators knowledge, there is no study that examined the effect of melatonin on inhaled isoflurane requirements intraoperatively. So, in this study, the effect of melatonin will be assessed on intraoperative inhaled isoflurane requirements in patients undergoing open nephrectomy under general anaesthesia by using entropy

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing nephrectomy under general anesthesia aged from 20 to 60 years.
* ASA 1 or 2.
* BMI 25 to 30

Exclusion Criteria:

* Patients with uncontrolled hypertension.
* Patients presenting with (IHD, significant arrhythmias, heart failure).
* Allergy to melatonin.
* History of epileptic seizures, psychoactive medications, neurological disorders or trauma.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-04-10 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Inhaled isoflurane requirement (volume%) to maintain entropy readings 40-60 | 2 hours
  Inhaled Isoflurane requirement (volume %) will be titrated to maintain state entropy (SE) and response entropy (RE) readings 40-60 measured using GE carestation 650-crescent pulse anaesthesia machine(6).

SECONDARY OUTCOMES:
Total morphine consumption over 24 hours postoperative | 24 hours
Total intraoperative fentanyl consumption | 2 hours
  The sum of fentanyl top up doses will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Amany Hassan Saleh, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No